CLINICAL TRIAL: NCT04063020
Title: Psychic Stakes of Reconstructive Plastic Surgery in Children With Ear Aplasia
Acronym: EPCHIRPRORL
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Other Study IDs: APHP190363; 2019-A00908-49 (Other: IDRCB number)
Record Dates: First submitted 2019-06-04; First posted 2019-08-20 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Ear Aplasia
Keywords: Ear aplasia; Reconstructive plastic surgery; Subjective experience; Psychic stakes; Psychodynamic evaluation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Reconstructive plastic surgery procedure: Minors with ear aplasia and initiating a reconstructive plastic surgery procedure
  Interventions: Behavioral: Psychological monitoring

INTERVENTIONS:
Behavioral: Psychological monitoring — Discussions with the psychologist PhD student before and after every surgery times : 3 discussions.
  * Before the first surgery (about 1 month before) Clinical interview Rorschach and TAT (Thematic Apperception Test) Drawing a person test Self Questionnaires : KIDSCREEN-27 and CDI Children's Depression Inventory- de Kovacs et Beck (1977)
  * Before the second surgery (3 months later the first surgery) Clinical interview Drawing a person
  * After the second surgery (15 months later the first surgery) Clinical interview Rorschach and TAT (Thematic Apperception Test) Drawing a person test Self Questionnaires : KIDSCREEN-27 and CDI Children's Depression Inventory- de Kovacs et Beck (1977)

SUMMARY:
The objective of the study is to analyse :

* Psychic experience of ear aplasia in children ;
* the modalities of their psychic functioning ;
* and the psychological repercussions of the plastic reconstruction surgery

DETAILED DESCRIPTION:
Children with an ear aplasia have various cares (ENT, speech therapy, hearing aids and tomodensiometry) up to the proposal of the plastic reconstruction surgery at 9/10 years old.

The surgical technique used and preferred within Necker Hospital for these children is that of Saturo Nagata (1994).

This surgical protocol takes place in two times, spaced by 9 months. This surgery does not allow hearing better since it targets is only a reconstruction of the pinna. To date, no research has highlighted the subjective experience of a child with an aplasia of ear and of what this surgery engages and demands on the side of psychological work.

The purpose of this research is to interrogate the children's subjective experience with an unilateral ear aplasia and who wishes a plastic reconstruction surgery for their aplase ear.

ELIGIBILITY:
Inclusion Criteria:

* Minors of 10 to 16 years old
* Unilateral ear aplasia with or without articulatory disorders, followed and engaged in reconstruction surgery procedure within the ENT service of cervico-facial surgery of the Necker Hospital
* Children wishing a plastic reconstruction surgery and having received the approval of the medical team
* Francophone children
* Holders of parental authority and child voluntary for the research

Exclusion Criteria:

* Illiterate children
* Severe intellectual deficit
* Bilateral aplasia
* Syndromic impairment

Ages: 10 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Minors with ear aplasia with or without articulatory disorders, without syndromic impairment and initiating a reconstructive plastic surgery procedure at Necker Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2020-01-18 (Actual); Primary Completion 2022-12-23 (Actual); Study Completion 2022-12-23 (Actual)

PRIMARY OUTCOMES:
Hermann Rorschach test | 1 year
  Hermann Rorschach test (1927) Test or projected test composed of 10 boards. Analysis by the psychogram (following the Chabert method).
  Psychic functioning of the child by description of: the mechanisms of defenses, the type of anxiety, the affective tone and the image of the body. The capacity to give adapted responses according to the boards as well as the narrative capacity of the child will make it possible to release tracks as for its psychic functioning.
Thematic Apperception Test | 1 year
  TAT: Thematic Apperception Test by MURRAY H.A. (1935) Projective test where the boards are different from the sex of the child (boy 13 boards, girls 14 boards).
  Quantitative analysis using the 4-dimensional tabulation sheet :
  * Series A: Rigidity
  * Series B: Lability
  * Series C: Conflict Avoidance
  * Series E: Emergencies of Primary Processes
  Psychic functioning of the child by description of: the mechanisms of defenses, the type of anxiety, the affective tone and the image of the body. The capacity to give adapted responses according to the boards as well as the narrative capacity of the child will make it possible to release tracks as for its psychic functioning.
Inventory of Childhood Depression | 1 year
  CDI: Inventory of Childhood Depression by M. Kovcas & A.T. Beck (1977) L.MOOR and C.MACK.
  Scale from 7 to 17 years. The score ranges from 0 to 54. The scale of rating goes from 0 to 2 with an alternation in the quotation of the articles so that the subject is not influenced by a same scheme of proposal by item.
  A score greater than or equal to 15 would be synonymous with depression but confirmed in clinical interview.
KIDSCREEN-27 | 1 year
  KIDSCREEN-27 from Kidscreen group europe (2006) -42 authors in all- The KIDSCREEN-27 is scored on a 5 point scale (1 = not at all, 2 = a little, 3 = moderately, 4 = a lot, 5 = extremely).
  Assessement of quality of life in children.
  The score can be calculated for each dimension:
  * Physical activities and health - 5 items;
  * The mood in general and the feeling - 7 elements;
  * Family life and free time - 7 articles;
  * Friends (social support and peers) - 4 elements;
  * At school (School Environment) - 4 elements.

CONTACTS AND LOCATIONS:
Overall Officials: Flora Aubertin, Psychologist, Principal Investigator — Assistance Publique - Hôpitaux de Paris; Françoise Denoyelle, MD, PhD, Study Director — Assistance Publique - Hôpitaux de Paris; Karinne Gueniche, Psychologist, Psychoanalyst, Study Director — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Necker-Enfants Malades, Paris, France

IPD SHARING:
Plan to Share IPD: No